CLINICAL TRIAL: NCT06804122
Title: Effects of Exercise-based Rehabilitation on Exercise Capacity, Quality of Life and Physical Activity in Patients With Pulmonary Artery Disease
Brief Title: Exercise-based Rehabilitation in Patients With Pulmonary Arterial Hypertension
Acronym: PAHexercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere Heart Hospital (Other)
Collaborators: Tampere University Hospital (Other); Tampere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R24101
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Exercise-based rehabilitation; Intervention
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Intervention Model Description: Exercise-based out-patients intervention is implemented to all particitpants who will undergo rehabiliation for pulmonary arterial hypertension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise-based outpatient rehabiliation (Experimental): All patients are allocated to this treatement arm where they are provided with structured guidance for implementation of exercise rehabiliation in an out-patient setting.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Patients are counseled how to do endurance training and strenght training at home by a trained physiotherapist.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare and severe disease characterized by elevation of pulmonary artery pressure (PAP) and increased pulmonary vascular resistance (PVR) due to the narrowing of small pulmonary arteries. The European Society of Cardiology (ESC) and the European Respiratory Society (ERS) recommend supervised exercise-based rehabilitation as part of the treatment of PAH patients alongside optimal medical therapy (Level of evidence A, Class of recommendation I).

Studies on exercise-based rehabilitation for PAH patients are limited, and most interventions have been conducted at least partially in hospital settings. Unlike more common cardiovascular diseases, there are no detailed international exercise guidelines tailored specifically for PAH patients.

This study aims to verify that a group-based outpatient rehabilitation protocol suitable for the Finnish healthcare system improves exercise capacity, quality of life, and physical activity of PAH patients and is safe for appropriately selected patients. Additionally, the study aims to determine whether PAH patients adhere to regular exercise training and whether physical activity increases in the long term.

The goal is to assess whether an outpatient rehabilitation protocol, designed for the Finnish healthcare system, can achieve similar results to those observed in previous international studies. The primary outcome measure is the change in the six-minute walking distance (6MWD) compared to the patient's baseline. Long-term 6MWD data are often available for patients. The 6MWD is the most commonly used primary outcome in randomized and controlled PAH drug trials, and improvements in this test have been the basis for drug approvals. An improvement of 33 meters in the 6MWD is considered clinically significant, and the goal is to achieve this change with group-based outpatient rehabilitation.

Secondary outcomes include changes in quality of life (SF-36), WHO functional class, NT-proBNP levels, echocardiographic parameters, ESC/ERS risk-stratification score (four-strata model), muscle strength, respiratory measures, balance, daily step count, and insomnia severity.

DETAILED DESCRIPTION:
Effects of group form exercise-based outpatient rehabilitation to Exercise Capacity, Quality of Life and Physical Activity in pulmonary artery hypertension (PAHexercise)

Pulmonary arterial hypertension (PAH) is a rare, severe and life-threatening disease with a poor prognosis, even with current medical treatments. In addition to medication, exercise rehabilitation has been shown to positively impact patients' functional capacity and quality of life. Following the diagnosis, patients often reduce their physical activity, experiencing hesitancy and uncertainty regarding safe exercise practices. However, the 2022 ESC/ERS international treatment guidelines recommend exercise rehabilitation for PAH patients with evidence level 1A. The strongest evidence for the benefits of rehabilitation comes from international multicenter studies, where rehabilitation has primarily occurred in hospital settings. There is no suitable or feasible guideline for outpatient-based exercise rehabilitation. However, studies indicate that exercise rehabilitation is safe for medically stable patients.

The aim of our research is to investigate and describe whether group-based outpatient exercise rehabilitation has an impact on the exercise capacity, quality of life, and physical activity of patients with pulmonary arterial hypertension. Additionally, we aim to develop an effective model for outpatient exercise rehabilitation for Finnish PAH patients. The rehabilitation will be supervised by experienced physiotherapists. Only patients in stable condition under effective medication will be included in the study, ensuring the safety of the rehabilitation. Furthermore, international safety standards, such as those related to oxygen saturation, heart rate, and hemoglobin levels, will be adhered to. Overexertion will be avoided. The rehabilitation sessions will take place in the facilities of the Tampere Heart Hospital, and a contingency plan has been developed to manage any adverse events.

Objectives, Primary, and Secondary Outcomes

The study aims to:

* Demonstrate the efficacy of a group-based outpatient rehabilitation program in improving the physical performance, quality of life, and physical activity of PAH patients.
* Assess long-term adherence to regular exercise training.
* Compare results to international standards to establish the program's suitability within the Finnish healthcare system.

Primary Outcome: Change in 6MWT results compared to baseline.

Secondary Outcomes:

* Change in Quality of life (SF-36).
* Change in WHO functional classification.
* Change in NT-proBNP biomarker levels.
* Changes in echocardiographic parameters.
* Change in the ESC risk classification score.
* Changes in muscle strength, respiratory parameters, balance, daily step count, and insomnia severity.

Research Methods

The study is a prospective, observational, non-controlled, quantitative study. It is a non-randomized case study focusing on a small group in a specific context. Quantitative methods will be used to analyze data, using participants' baseline and historical follow-up results as comparators.

Due to the small patient cohort, a formal power analysis is not feasible. However, the goal is to demonstrate that the chosen rehabilitation method achieves a median improvement in 6MWT results comparable to those observed in large, randomized multicenter trials.

Schedule of the Research

Participants (maximum 20, minimum 8) will be recruited between 2025 and 2030. PAH is a rare disease, with international studies including sample sizes ranging from 7 to 183 participants.

The target group comprises PAH patients under follow-up at the cardiology outpatient clinic of Tays Heart Hospital.

Implementation of the Research

Inclusion and Exclusion Criteria

Inclusion Criteria:

* Adults over 18 years old residing in Tampere or nearby municipalities.
* WHO functional classification II-III.
* Commitment to the exercise program.
* Stable disease condition with no PAH medication changes in the two months prior.
* No recent syncope or arrhythmias causing symptoms within the past two months.

Exclusion Criteria:

* Severe pulmonary disease or left ventricular failure (HFrEF).
* Pregnancy.
* Severe congenital heart defect (Eisenmenger syndrome).
* Severe liver disease.
* Acute inflammatory condition.
* Severe anemia (hemoglobin ≤ 75% of the lower reference limit).
* Systolic blood pressure below 85 mmHg.
* Recent syncope.
* Other significant conditions affecting physical capacity, such as severe neurological diseases or musculoskeletal issues.
* Untreated severe arrhythmias.
* Changes in PAH medication during the rehabilitation program.

Execution of Rehabilitation The program includes once a week total 15 group exercise sessions led by a physiotherapist, along with three individual sessions for baseline, post-program, and one-year follow-up assessments. Group sizes are limited to a maximum of four participants.

Each session consists of:

1. Warm-up.
2. Circuit training focusing on muscle strength.
3. Cool-down. Participants will also follow a home-based exercise program, including endurance, strength, and respiratory exercises.

Metrics Performance metrics include the 6MWT, grip strength, chair stand test (10 repetitions), single-leg standing, respiratory function tests, and inspiratory muscle strength measurements. Participants will complete the SF-36, ISI (Insomnia Severity Index), and IPAQ (International Physical Activity Questionnaire) surveys before, after, and one year after the program. Daily physical activity will be tracked using a step counter.

Echocardiographic evaluations will be conducted before and after the program, with potential mid-program assessments. Blood tests will monitor NT-proBNP and hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old residing in Tampere or nearby municipalities.
* WHO functional classification II-III.
* Commitment to the exercise program.
* Stable disease condition with no PAH medication changes in the two months prior.
* No recent syncope or arrhythmias causing symptoms within the past two months.

Exclusion Criteria:

* Severe pulmonary disease or left ventricular failure (HFrEF).
* Pregnancy.
* Severe congenital heart defect (Eisenmenger syndrome).
* Severe liver disease.
* Acute inflammatory condition.
* Severe anemia (hemoglobin ≤ 75% of the lower reference limit).
* Systolic blood pressure below 85 mmHg.
* Recent syncope.
* Other significant conditions affecting physical capacity, such as severe neurological diseases or musculoskeletal issues.
* Untreated severe arrhythmias.
* Changes in PAH medication during the rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in six-minute walking test result | 12 weeks
  Each participant performs a six-minute walking test at baseline (before exercise-based intervention) and after the intervention that lasts 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jussi A Hernesniemi, MD PhD, Study Chair — Tampere Heart Hospital
Locations (1):
- Tampere Heart Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
Due to Finnish legislation, IPD cannot be shared outside the European Union. However, upon reasonable request the data can be shared for scientific purposes pending the approval of the study board